CLINICAL TRIAL: NCT05992272
Title: Cue Effects in Human Addiction: Pavlovian to Instrumental Transfer
Acronym: ReCoDe
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Andreas Heinz, head of Department of Psychiatry and Psychotherapy | CCM, principle investigator, Charite University, Berlin, Germany
Other Study IDs: 402170461
Record Dates: First submitted 2023-06-30; First posted 2023-08-15 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use Disorder (AUD); Alcoholism; Substance Use Disorders; Smoking, Tobacco; Stress Reaction; Stress
Keywords: substance use disorder (SUD), cognitive control/interference; alcohol use disorder (AUD); Smokers; general and outcome-specific Pavlovian to instrumental transfer; chronic and acute stress; Amygdala; Stroop Test; Ventral Striatum; Neuroimaging; Humans; Surveys and Questionnaires; Reward; Fractals; Cues
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Tobacco Smoking; Fractures, Stress; Bronchiolitis Obliterans Syndrome | interventions — Psychological Tests; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- alcohol use disorder (AUD): Participants with alcohol use disorder (mild to moderate or severe if no withdrawal symptoms) including:
  * daily smokers (at least 1 cigarette per day in last 3 months)
  * non-daily (min 1x/last 3months)
  * non-smokers
  Interventions: Biological: fMRI imaging (BOLD); Biological: sMRI (structure); Behavioral: Trier Social Stress Test; Behavioral: PIT paradigm; Behavioral: Counting Stroop task; Behavioral: No-go Simon task; Diagnostic Test: Stop Signal Task; Diagnostic Test: blood samples; Diagnostic Test: questionnaires for chronic stress; Diagnostic Test: hair samples; Diagnostic Test: saliva samples; Diagnostic Test: EMA assessment; Diagnostic Test: clinical diagnostic
- non-AUD: Participants with a maximum of 1 AUD criteria according to DSM-5, including:
  * daily smokers (at least 1 cigarette per day in last 3 months)
  * non-daily (min 1x/last 3months)
  * non-smokers
  Interventions: Biological: fMRI imaging (BOLD); Biological: sMRI (structure); Behavioral: Trier Social Stress Test; Behavioral: PIT paradigm; Behavioral: Counting Stroop task; Behavioral: No-go Simon task; Diagnostic Test: Stop Signal Task; Diagnostic Test: blood samples; Diagnostic Test: questionnaires for chronic stress; Diagnostic Test: hair samples; Diagnostic Test: saliva samples; Diagnostic Test: clinical diagnostic

INTERVENTIONS:
Biological: fMRI imaging (BOLD) — Will be used to investigate neural correlates of PIT effects by measuring the blood oxygenation level dependent (BOLD) response of neural activation in the mesolimbic system.
Biological: sMRI (structure) — Will be used to investigate neural correlates of PIT effects by identifying abnormalities in cortical gray and white matter volume.
Behavioral: Trier Social Stress Test — Will be used to assess the effect of acute stress induction on behavioral and neural PIT effects. The induced stress is generated in a social context, where the participants are asked to prepare a job interview for their dream job and to present it in front of a three-member jury.
Behavioral: PIT paradigm — The paradigm consists of four parts:
  In the first part, an instrumental learning task is completed in which subjects must learn which stimuli require a response and which do not. In the second part, a classical (Pavlovian) conditioning task is then completed in which subjects learn by passive viewing which stimuli are associated with certain amounts of money. The third part measures to which instrumental responses (learned in Part 1) are modulated by the presentation of the classically conditioned stimuli (learned in Part 2). At the same time drug-associated stimuli are presented in the background measuring to which extent they conflict with the learned instrumental behavior. In the last part, query trials are implemented in which the participants have to choose between two pictures to assess the relative cue value.
Behavioral: Counting Stroop task — Will be used to assess interference at stimulus level. Here either one, two, three or four identical digits from 1 to 4 are shown. Number and denotation of digits are either congruent (1, 22, 333, 4444; 88 trials) or incongruent (111, 2222, 3, 4444; 88 trials). Subjects have to indicate how many digits were shown
Behavioral: No-go Simon task — Will be used to measure interference at the response level and response inhibition. We will show arrows either pointing to the left or right. The arrow can either be shown on the left or the right side of the display. In congruent trials, direction and position are the same, whereas they differ in incongruent trials. Participants have to indicate the direction of the arrow and ignore the position.
Diagnostic Test: Stop Signal Task — Will be used to examine inhibitory control. The participants tap the left and right side of the screen to smash two falling fruits. When the fruits pass two circles, subjects are required to tap both sides of the screen. In "stop trials" one of the fruits turns brown (rotten), indicating the corresponding side of the screen should not be tapped.
Diagnostic Test: blood samples — for genetic and epigenetic testing, especially for exploratory outcome prediction using polygenic risk scores.
Diagnostic Test: questionnaires for chronic stress — * Perceived Stress Scale
  * Social Readjustment Rating Scale
  * Trier Inventory for the Assessment of Chronic
Diagnostic Test: hair samples — Hair cortisol measurement (3 cm hair segments) will be used to assess chronic stress.
Diagnostic Test: saliva samples — Assessing acute stress effects in AUD.
Diagnostic Test: EMA assessment — We will use smartphones with additional mobile sensors (wearables), which will be used to measure physical activity, data on location (GPS), geolocation-based triggering of e-Diaries, self-reported stress reactivity, cue exposure (encounters with drug-related stimuli in real life), drug craving, impulsivity and drug consumption (priming doses, binges and continuous use of all drugs of abuse).
  Groups: alcohol use disorder (AUD)
Diagnostic Test: clinical diagnostic — SKID-I Interview neurocognitive and psychopathological testing

SUMMARY:
Individuals with substance use disorders (SUD) have to cope with drug-related cues and contexts, which can affect instrumental drug seeking as shown with Pavlovian to instrumental transfer (PIT) paradigms in animals and humans. The investigators aimed to investigate the impact of acute and chronic stress on Pavlovian-to-instrumental transfer (PIT), how PIT it is associated with cognitive control abilities and whether such effects predict losing vs. regaining control in subjects with AUD. Moreover, the investigators aimed to develop a novel full transfer task that assesses both, general and specific PIT to investigate whether specific PIT differs between alcohol use disorder (AUD) and control subjects.

DETAILED DESCRIPTION:
This project has four research aims:

1. The investigators want to assess the effects of acute as well as repeated stress exposure on PIT and its neuroimaging correlates, and the investigators will test whether modulation of PIT by stress predicts losing vs. regaining control of drug intake in mild to moderate AUD subjects.
2. The investigators will investigate how cognitive control abilities (e.g. interference control and response inhibition) are related to the costs of interference between Pavlovian and instrumental control in PIT.
3. The investigators will compare PIT, its relation to cognitive control, and the neural mechanisms between different drugs of abuse by investigating participants with AUD and also smokers.
4. The investigators will develop an outcome-specific PIT paradigm with alternative (food) and drug rewards to compare AUD and healthy controls, and the investigators will explore communalities and differences in behavioral and neural processes between general PIT and outcome-specific PIT.

Therefore, the investigators conduct 3 Experiments with the following Hypotheses:

Experiment 1:

Here the investigators assess on a behavioral and neural level a general PIT task that consists of four parts:

In the instrumental part, participants have to learn which shells to collect or leave in order to gain as much money as possible; the correct choice is probabilistically rewarded in 80% of all times. Absolutely unrelated to this instrumental part, during Pavlovian conditioning colorful fractals are presented in the back of the screen, which have been passively paired either with monetary gain, no change or monetary loss, i.e. they act as positively valued, neutral or negatively valued cues. These fractals thus act as independent, Pavlovian conditioned background stimuli and interact with instrumental behavior in the unrelated third transfer part of the PIT task. Also, the investigators assess the effects of drug-specific cues in the background on instrumental behavior during this transfer part. To avoid further learning, the transfer part will be conducted under nominal extinction. Finally, query trials, in which participants will have to choose one of two pictures will to assess the relative cue value.

Acute stress will be induced by the Trier Social Stress Test (TSST), chronic stress will be assessed by questionnaires and hair cortisol.

Hypothesis 1a:

Acute and chronic stress exposure increase behavioral and neural PIT effects elicited by monetary Pavlovian conditioned stimuli (CS) and decrease inhibitory effects of alcohol Pavlovian CS. Functional correlates of PIT effects will be found in the amygdala and in the ventral striatum.

Hypothesis 1b:

Following stress exposure, high PIT effects elicited by monetary Pavlovian CS and low inhibitory effects elicited by alcohol Pavlovian CS predict higher subsequent alcohol intake in the follow-up period of 6 months.

Methods:

Between group analysis: The investigators will analyze on a behavioral and imaging level how acutely consuming AUD subjects and matched controls differ regarding money- and alcohol-related PIT.

Within-group analysis: The investigators will analyze how acute stress affects PIT effects. This 2x2 design (1 within-group subject factor with two levels: STRESS vs. NO STRESS and 1 between-group subject factor with two levels: AUD vs. matched controls) will be tested on a behavioral and neural level.

Experiment 2:

In this experiment, the investigators will utilize a 2x3 factorial group design. Participants will be categorized into two main groups: those with AUD and those without (non-AUD). Each of these groups will be further divided into three subgroups: daily smokers, non-daily smokers and non-smokers. Each cell (individual subgroup) will consist of 35 subjects. In addition to the PIT task described above, the N = 210 participants will additionally perform a Counting Stroop task and a No-go Simon task. Participants will also perform a stop signal task during functional MRI (fMRI).

Methods:

Interference Costs: Interference costs will be calculated based on error rate (ER) and reaction time (RT) differences between task conditions, e.g., incongruent vs. congruent conditions.

Between-group analysis: the investigators will examine group differences in the interference PIT effect at both the behavioral and neural levels using a two (AUD vs. non-AUD) by three (daily smokers vs. non-daily smokers vs. non-smokers) design. In addition, the investigators aim to investigate the associations between the interference PIT effect and other continuous measures: Alcohol Use Disorders Identification Test (AUDIT), Fagerström Test for Nicotine Dependence (FTND), along with quantity-frequency indices.

Other analysis: In order to gain a better understanding of the mechanisms underlying PIT, the investigators will also fit a drift diffusion model to the behavioral data and explore the connectivity within the neural networks during PIT in relation to the connectivity during the stop signal task (response inhibition).

Hypothesis 2a:

Interference costs (i.e. increased error rate [ER] in instrumental responses) during PIT are associated with interference costs at the stimulus level (Stroop task) and at the response level (No-go Simon task), and these costs will also be correlated with the ER during response inhibition (No-go Simon task).

Hypothesis 2b:

The investigators hypothesize that the interference PIT effect will be more pronounced in the AUD group compared to the non-AUD group. The investigators also anticipate that the effect will be stronger in the smoker group. Furthermore, the investigators hypothesize a positive correlation between the PIT effect and AUDIT, FTND scores, as well as the quantity and frequency of use. As the behavioral PIT effect intensifies, the investigators expect corresponding neural responses to similarly increase.

Experiment 3:

The investigators here use a newly-developed full PIT paradigm that introduces primary reinforcers, i.e. alcoholic and soft drinks (that the investigators administer on a trial-by-trial basis). Furthermore, the investigators implemented additional Pavlovian stimuli to examine both general and outcome-specific PIT effects. General PIT effects occur when positively valued environmental Pavlovian stimuli enhance instrumental responding regardless of the reinforcer being used. Here, stimuli that are associated with e.g. monetary rewards can enhance instrumental responding for alcohol drinks, demonstrating a general motivational effect. In contrast, during outcome-specific PIT, this effect is limited for the same stimulus-reward association. For instance, Pavlovian stimuli associated with a soft drink promote choices for the same soft drink outcome only.

Methods:

Between-group Analysis: The investigators will assess the outcome-specific PIT effects by measuring the change in the proportion of alcohol choices when the alcohol cue is presented versus when the soft drink (juice) cue is shown. On the other hand, the investigators will define general PIT effects as the increase in button presses (i.e., slope) corresponding to the increased valence of the conditioned monetary cues. The investigators plan to examine the differences in both specific and general PIT effects at both the behavioral and neural levels between the AUD group and the non-AUD group, controlling for smoking status. Additionally, the investigators will investigate the relationship between specific and general PIT effects and AUDIT, along with quantity-frequency measures Comparison between the two PIT tasks: the investigators will explore similarities and differences in PIT effects between the full PIT paradigm and the previously-mentioned single-lever PIT paradigm.

Stress: the investigators will test whether levels of chronic stress (assessed with questionnaires and hair cortisol as for Experiment 1) moderate outcome-specific and full PIT effects.

Hypothesis 3a:

The investigators expect that both outcome-specific and general PIT effects will be stronger in participants with AUD compared to those without AUD, evident at both behavioral and neural levels. Additionally, the investigators predict positive associations between PIT effects and both AUDIT scores and quantity-frequency measures.

Hypothesis 3b:

the investigators hypothesize that the PIT effect found in the single-lever PIT task is more strongly associated with the general PIT and less strongly associated with the outcome-specific PIT effect in the full PIT task.

Hypothesis 3c:

Increased chronic stress will enhance effects of both general and outcome-specific PIT.

ELIGIBILITY:
Inclusion Criteria:

* males and females between 16-65 years of age
* AUD subjects only: meet a minimum of 2 criteria for DSM-5 alcohol-related disorder (AUD) (not requiring withdrawal as assessed by an independent psychiatrist) and AUDIT > 4
* Smokers: Daily smokers only: smoke 7 days/week during the last three months
* Non-daily smokers only: smoke at least once but less than 7 days/week during the last three months
* Ability to consent to the study and complete the questionnaires
* Sufficient language skills: German
* Availability between 3pm-6pm on 2 consecutive days (Experiment 1, acute stress question)
* Females only: luteal phase (Experiment 1, acute stress question)

Exclusion Criteria:

* Lifetime diagnosis according to DMS-5 for: Bipolar disorder, schizophrenia, schizophrenia spectrum disorder, substance dependence except for alcohol, nicotine, or cannabis
* Currently meeting DSM-5 diagnostic criteria for a depressive episode, suicidal ideation
* Past traumatic brain injury or severe neurological disease (such as dementia, Parkinson's disease, multiple sclerosis)
* Pregnancy or breastfeeding
* Ingestion of medications known to interact with the CNS in the 10-day period prior to study participation or less than 4 half-lives after last ingestion (rapid urine test)
* MR contraindications (e.g., pacemakers, metallic or electronic implants, metallic splinters, surgical staples)
* Color vision deficiency
* Sensorineural hearing loss of 30 dB or greater,
* Tinnitus
* Presence of claustrophobia
* Acute alcohol intoxication at MRI appointments verified by breath alcohol testing or drug intoxication verified by rapid urine testing
* For women only: not peri- or postmenopausal, not taking contraceptives (Experiment 1, acute stress question)

Ages: 16 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All groups will be recruited from general population via advertisement (e.g. ebay Kleinanzeigen, Facebook) and notes (e.g. blackbords, intranet) in Berlin and Dresden
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Neural PIT effect day 1 | Day 1
  blood oxygenation level dependent (BOLD) response, investigation of neuronal activation of the mesolimbic system in AUD patients and controls using 3 Tesla magnetic resonance imaging following Stress or Placebo intervention OR no intervention
Neural PIT effect day 2 | Day 2
  a subsample of subjects has a second assessment with blood oxygenation level dependent (BOLD) response, investigation of neuronal activation of the mesolimbic system in AUD patients and controls using 3 Tesla magnetic resonance imaging following Stress or Placebo intervention
Behavioral PIT effect on performance day 1 | Day 1
  strength of PIT effect assessed with the PIT paradigm. Performance (correct choices) will be recorded. Stronger PIT effects are associated with higher performance (percent correct choices) in congruent versus lower performance in incongruent trials.
Behavioral PIT effect on velocity day 1 | Day 1
  strength of PIT effect assessed with the PIT paradigm. Velocity will be recorded. Stronger PIT effects are associated with higher velocity in conditions with positively valued background stimuli and lower velocity with negatively valued background stimuli.
Behavioral PIT effect on velocity day 2 | Day 2
  a subsample of subjects has a second assessment with the PIT paradigm (parallel version) following Stress or Placebo intervention. At this second day the investigators calculate velocity PIT effect only.
Chronic stress effects on hair cortisol in picogram/milligram | retrospective assessment before PIT testing at Day 1
  chronic stress assessment via:
  - hair cortisol measurement (3 cm hair segments)
Chronic stress quenstionnaire 1 | retrospective assessment before PIT testing at Day 1
  chronic stress assessment via:
  - Trier Inventory for the Assessment of Chronic Stress (TICS; assessing chronic stress over the last three months, likert scale 0-4, with zero meaning never and four meaning very often; high values stand for more stress))
Chronic stress quenstionnaire 2 | retrospective assessment before PIT testing at Day 1
  chronic stress assessment via:
  - Social Readjustment Rating Scale (SRRS; assessing chronic stress life events of the last year, scaling asking for yes or no. higher values represent more stressful live events over the last year)
Chronic stress quenstionnaire 3 | retrospective assessment before PIT testing at Day 1
  chronic stress assessment via:
  - Perceived Stress Scale (PSS; assessing chronic stress over the last month, likert scale 0-4, with zero meaning never and four meaning very often; high values stand for higher perceived stress)
cognitive control Stroop effect | Day 1
  Cognitive control assessment via:
  - Counting Stroop task
cognitive control Simon effect | Day 1
  Cognitive control assessment via:
  No-go Simon task
cognitive control interference effect | Day 1
  Cognitive control assessment via:
  Stop Signal reaction time task
Acute stress day 1 | Day 1
  Acute stress inducting using:
  Trier social stress test (TSST) OR placebo (randomized across days between subjects)
Acute stress day 2 | Day 2
  Acute stress inducting using:
  Trier social stress test (TSST) OR placebo (randomized across days between subjects)

SECONDARY OUTCOMES:
Saliva cortisol concentration in nmol/litre | Assessment before, during and after TSST (-60 minutes, 0 minutes, +10 minutes, +20 minutes, +30 minutes,+ 50 minutes, +80 minutes)
  Acute stress effects in AUD and HC
alcohol consumption after 12 months | 12 months after testing for behavioral and neural PIT effects
  alcohol drinking amount (quantity, frequency) during a follow-up period of 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Charite - Universitätsmedizin Berlin, Berlin
  - Technische Universität Dresden, Dresden

REFERENCES:
- [Result] Belanger MJ, Chen H, Hentschel A, Garbusow M, Ebrahimi C, Knorr FG, Zech HG, Pilhatsch M, Heinz A, Smolka MN. Development of Novel Tasks to Assess Outcome-Specific and General Pavlovian-to-Instrumental Transfer in Humans. Neuropsychobiology. 2022;81(5):370-386. doi: 10.1159/000526774. Epub 2022 Nov 14. PMID 36380640